CLINICAL TRIAL: NCT04202276
Title: The Study of Nutrition of Children and Adolescents With GERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Responsible Party: Principal Investigator, Sergey Morozov, Leading researcher, Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: AAAA-А19-119041090031-7
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: GERD in Children; GERD
Keywords: gastroesophageal reflux; weight; obesity; nutrition; GERD; esophageal pH-impedance; food frequency questionnair
MeSH Terms: conditions — Gastroesophageal Reflux; Body Weight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with GERD (Other): The data of Food frequency questionnaire (FFQ), 24-hours oesophageal pH-impedance examination, GERD-Q questionnaire to be performed in children and adolescents with GERD.
  Interventions: Other: diet assessment
- Control group (Other): The same examinations as in experimental group are to be performed in patients of the control group (no GERD according to the results of the examination): Food frequency questionnaire (FFQ), 24-hours oesophageal pH-impedance examination, GERD-Q questionnaire.
  Interventions: Other: diet assessment

INTERVENTIONS:
Other: diet assessment — Food frequency questionnaire to investigate differences in diet of children and adolescents with GERD compared to the age- and sex matched control group.

SUMMARY:
This trial is to study the aspects of nutrition in children and adolescents with GERD compared to the sex and age-matched control group

DETAILED DESCRIPTION:
The aim of the study is to assess the differences in nutrition of pediatric patients with GERD compared to the control group. The secondary aim is to study possible associations of the data on nutritional habits revealed with the use of food frequency questionnaire (FFQ) and the data of 24-hours oesophageal pH-impedance examination.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate (written informed consent and consent from parents or legal representative according to the local law);
* Age 6 to 17 years old inclusive,
* Possibility to assess symptoms, data of the medical history and receive answers to the questions about usual diet.

Exclusion Criteria:

* history of abdominal surgery;
* presence of varicose veins of the stomach and/or the oesophagus either in medical history or found during the study;
* inability to tolerate at least one of the invasive procedures or lacking data of the other instrumental examinations required by protocol;
* general condition of the patient making impossible to perform all the examinations or when performing the procedures is not safe and reasonable based on the opinion of the investigator that it may exacerbate the disease flow or put the patient at risk;
* intake of medications which may influence the clinical and instrumental data, including, but not limited to: non-steroid anti-inflammatory agents, glucocorticosteroids (except for skin products, if they were used for 2 weeks or less at the time of inclusion into the study), medications affecting adrenergic, acetylcholine receptors, antidepressants, tranquillizers, sedatives, those with known local irritant effect on the gastrointestinal tract mucosa; the use of proton pump inhibitors and H2 receptors blockers are not allowed during the study, a wash-out period for at least 2 weeks is necessary before the enrolment.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Energy value of the ration | An average of 1 year
  value of mean daily consumption of the energy by food frequency questionnaire, kcal/day
total fat consumption | An average of 1 year
  value of mean daily consumption of fats by food frequency questionnaire, G/day
total carbohydrate consumption | An average of 1 year
  value of mean daily consumption of carbohydrates, by food frequency questionnaire, G/day
total protein consumption | An average of 1 year
  value of mean daily consumption of protein by food frequency questionnaire, G/day
Dietary fibre consumption | An average of 1 year
  value of mean daily consumption of dietary fibre, by food frequency questionnaire, G/day

SECONDARY OUTCOMES:
Total number of gastroesophageal refluxes | 24-hours
  This measure is to be obtained by 24-hours oesophageal pH-impedance study
Number of acid gastroesophageal refluxes | 24-hours
  This measure is to be obtained by 24-hours oesophageal pH-impedance study
Number of weak-acid gastroesophageal refluxes | 24-hours
  This measure is to be obtained by 24-hours oesophageal pH-impedance study
Number of high gastroesophageal refluxes | 24-hours
  This measure is to be obtained by 24-hours oesophageal pH-impedance study
Acid exposure time | 24-hours
  This measure is to be obtained by 24-hours oesophageal pH-impedance study

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy B Nikityuk, Professor, Study Director — Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology; Tatiana Strokova, Professor, Study Chair — Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Locations (1):
- Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared by the request. No personal data of the participants is a subject for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: upon study completion. Available for 2 years according to the local low
Access Criteria: by request
URL: http://rosrid.ru

REFERENCES:
- [Derived] Borodina G, Morozov S. Children With Gastroesophageal Reflux Disease Consume More Calories and Fat Compared to Controls of Same Weight and Age. J Pediatr Gastroenterol Nutr. 2020 Jun;70(6):808-814. doi: 10.1097/MPG.0000000000002652. PMID 32443037